CLINICAL TRIAL: NCT05678257
Title: A Randomised, Open-label, Phase II, Dose/Schedule Optimisation Study of NUC-3373/Leucovorin/Irinotecan Plus Bevacizumab (NUFIRI-bev) Versus 5-FU/Leucovorin/Irinotecan Plus Bevacizumab (FOLFIRI-bev) for the Treatment of Patients With Previously Treated Unresectable Metastatic Colorectal Cancer
Brief Title: A Study of NUC-3373 in Combination With Other Agents in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A pre-planned initial analysis concluded that the study was unlikely to achieve its primary objective of demonstrating superior progression-free survival. Based on the Steering Committee's recommendation, the Sponsor has closed the study.
Sponsor: NuCana plc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NuTide:323; 2022-001459-17 (EudraCT Number)
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenocarcinoma; Colorectal Cancer Metastatic; Neoplasm, Colorectal
Keywords: Relapsed metastatic adenocarcinoma of colon/rectum; NUC-3373; Fosifloxuridine nafalbenamide; Leucovorin; Irinotecan; Bevacizumab; Antineoplastic agents; Chemotherapy; Second-line chemotherapy; Locally advanced cancer; Metastatic cancer; Neoplasm; 5-FU
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Leucovorin; Irinotecan; Bevacizumab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NUFIRI-bev on a Q1W NUC-3373 schedule (Experimental): Arm A: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
     * 90 minutes for the first dose
     * 60 minutes for the second dose (if first dose is tolerated)
     * 30 minutes for subsequent doses (if second dose is tolerated)
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1, 8, 15, and 22.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. NUC-3373 1500 mg/m2 over 120 minutes on Days 1, 8, 15, and 22.
  Interventions: Drug: Fosifloxuridine Nafalbenamide; Drug: Leucovorin; Drug: Irinotecan; Biological: Bevacizumab
- NUFIRI-bev on a Q2W NUC-3373 schedule (Experimental): Arm B: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
     * 90 minutes for the first dose
     * 60 minutes for the second dose (if first dose is tolerated)
     * 30 minutes for subsequent doses (if second dose is tolerated)
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1 and 15.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. NUC-3373 1500 mg/m2 over 120 minutes on Days 1 and 15.
  Interventions: Drug: Fosifloxuridine Nafalbenamide; Drug: Leucovorin; Drug: Irinotecan; Biological: Bevacizumab
- FOLFIRI-bev on a Q2W schedule (Active Comparator): Arm C: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
     * 90 minutes for the first dose
     * 60 minutes for the second dose (if first dose is tolerated)
     * 30 minutes for subsequent doses (if second dose is tolerated)
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1 and 15.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. 5-FU 400 mg/m2 bolus on Days 1 and 15.
  5. 5-FU 2400 mg/m2 infusion over 46 hours on Days 1 and 15.
  Interventions: Drug: Leucovorin; Drug: Irinotecan; Biological: Bevacizumab; Drug: 5-FU

INTERVENTIONS:
Drug: Fosifloxuridine Nafalbenamide — Intravenous infusion
  Other Names: NUC-3373; Nucleotide analogue
  Arms: NUFIRI-bev on a Q1W NUC-3373 schedule; NUFIRI-bev on a Q2W NUC-3373 schedule
Drug: Leucovorin — Intravenous infusion
  Other Names: Folinic acid; LV
Drug: Irinotecan — Intravenous infusion
  Other Names: Campto; Camptosar
Biological: Bevacizumab — Intravenous infusion
  Other Names: Avastin; Zirabev
Drug: 5-FU — Intravenous infusion
  Other Names: 5FU; 5-fluorouracil; Fluorouracil
  Arms: FOLFIRI-bev on a Q2W schedule

SUMMARY:
This is a randomized, open-label, dose/schedule optimization study comparing NUC-3373/leucovorin (LV)/irinotecan plus bevacizumab (NUFIRI-bev) to 5-FU/LV/irinotecan plus bevacizumab (FOLFIRI-bev) for the treatment of patients with unresectable metastatic colorectal cancer.

A total of 171 patients will be randomized 1:1:1 to either NUFIRI-bev on a weekly NUC-3373 schedule, NUFIRI-bev based on an alternate weekly NUC-3373 schedule, or FOLFIRI bev on an alternate weekly schedule. The main objectives are to assess and compare the efficacy and safety of the 3 regimens. Pharmacokinetics will be assessed on the 2 NUFIRI arms.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Histological or cytological confirmation of colorectal adenocarcinoma (excluding appendiceal and anal canal cancers, as well as signet-ring cell carcinoma) that is unresectable and metastatic.
3. Measurable disease (as defined by RECIST v1.1).
4. Received ≥2 months of a first-line fluoropyrimidine and oxaliplatin-containing regimen for metastatic disease or relapsed within 6 months of completing a fluoropyrimidine and oxaliplatin-containing neoadjuvant/adjuvant therapy. Previous treatment with standard of care chemotherapy regimens in combination with molecular targeted therapies (e.g., VEGF and EGFR pathway inhibitors and immuno-oncology agents) is permitted. Previous treatment with maintenance therapy (e.g., capecitabine) is also allowed. Patients who started on a fluoropyrimidine and oxaliplatin-containing regimen in any setting but must discontinue the oxaliplatin due to.toxicity or allergy (and are now unable to receive oxaliplatin) are considered eligible regardless of the number of cycles of oxaliplatin they received.
5. Known RAS and BRAF status. Patients with wild-type RAS tumours must have received prior treatment with an EGFR inhibitor, unless this was not standard of care according to relevant region-specific treatment recommendations.
6. Known UGT1A1 status, or patient consents to UGT1A1 status testing if unknown.
7. Known DPD activity status, or patient consents to DPD status testing if unknown. See exclusion criterion 1.
8. Age ≥18 years.
9. Minimum life expectancy of ≥12 weeks.
10. Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1.
11. Adequate bone marrow function as defined by: absolute neutrophil count (ANC) ≥1.5 × 109/L, platelet count ≥100 × 109/L, and haemoglobin ≥9 g/dL. Patients with benign neutropenia may be discussed on a case-by-case basis with the medical monitor.
12. Adequate liver function, as defined by: serum total bilirubin ≤1.5 × ULN), AST and ALT ≤2.5 × ULN (or ≤5 × ULN if liver metastases are present).
13. Adequate renal function assessed as serum creatinine <1.5 × ULN and glomerular filtration rate ≥50 mL/min (calculated by the Cockcroft-Gault method).
14. Serum albumin ≥3 g/dL.
15. Ability to comply with protocol requirements.
16. Female patients of child-bearing potential must have a negative serum pregnancy test within 7 days prior to the first study drug administration. This criterion does not apply to patients who have had a previous hysterectomy or bilateral oophorectomy. Male patients and female patients of child-bearing potential must agree to practice true abstinence (defined in Section 10.3.1) or to use two forms of contraception, one of which must be highly effective. These forms of contraception must be used from the time of signing consent, throughout the treatment period, and for 6 months following the last dose of any study medication. Oral or injectable contraceptive agents cannot be the sole method of contraception
17. Patients must have been advised to take measures to avoid or minimize exposure of the skin and eyes to UV light, including avoiding sunbathing and solarium use, for the duration of study participation and for a period of 4 weeks following the last dose of study medication

Exclusion Criteria:

1. History of hypersensitivity or current contra-indications to 5-FU, FUDR, or capecitabine.
2. History of hypersensitivity or current contra-indication to any of the combination agents required for the study.
3. History of allergic reactions attributed to components of the NUC-3373 drug product formulation.
4. History of hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies.
5. History of or known central nervous system or leptomeningeal metastases.
6. Symptomatic ascites, ascites currently requiring drainage procedures or ascites requiring drainage over the prior 3 months.
7. Mutant BRAF V600E status.
8. MSI high or dMMR.
9. Prior treatment with irinotecan.
10. Chemotherapy, hormonal therapy, radiotherapy (other than a short cycle of palliative radiotherapy [e.g., for bone pain]*), immunotherapy, biological agents, or exposure to another investigational agent within 21 days (or four times the half-life for molecular targeted agents, whichever is shorter) of first administration of study treatment:
11. Residual toxicities from prior chemotherapy or radiotherapy which have not regressed to Grade ≤1 severity (CTCAE v5.0), except for alopecia and residual Grade 2 neuropathy.
12. History of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, surgically excised or potentially curatively treated ductal carcinoma in situ of the breast, or low-grade prostate cancer or patients after prostatectomy. Patients with previous invasive cancers are eligible if treatment was completed >3 years prior to initiating the current study treatment, and the patient has had no evidence or recurrence since then.
13. Presence of an active bacterial or viral infection (including SARS-CoV-2, Herpes Zoster, Varicella Zoster or chickenpox), known Human Immunodeficiency Virus (HIV) positive or known active hepatitis B or C.
14. Presence of any uncontrolled concurrent serious illness, medical condition or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's ability to participate in the study or with the interpretation of the results (refer to protocol for further details).
15. Any condition that, in the judgment of the Investigator, may affect the patient's ability to provide informed consent and undergo study procedures.
16. Patients with a history of haemoptysis (1/2 teaspoon or more of red blood) within 6 months prior to enrolment.
17. Wound healing complications or surgery within 28 days of starting bevacizumab (wound healing must have been fully completed before starting bevacizumab). Investigators may allow patients to initiate treatment with the other study drugs (i.e., NUC-3373/5-FU, LV and irinotecan) on C1D1 but withhold bevacizumab for at least 15 days, but no longer than 28 days, to allow completion of wound healing in patients who would otherwise be eligible for the study, in line with standard local practice and after discussion with the Medical Monitor. Patients who have not received bevacizumab by C2D1 must be replaced.
18. Unhealed wound, active gastric or duodenal ulcer, or bone fracture.
19. Serious thromboembolic event in the 6 months before inclusion.
20. Patients with a history of haemorrhage within 6 months prior to enrolment.
21. Known inherited or acquired bleeding disorders.
22. Red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening.
23. Uncontrolled hypertension.
24. Severe proteinuria or nephrotic syndrome.
25. Acute intestinal obstruction or sub-obstruction, history of inflammatory intestinal disease or extended resection of the small intestine. Presence of a colic prosthesis.
26. History of abdominal fistulas, trachea-oesophageal fistulas, any other Grade 4 gastrointestinal perforations, non-gastrointestinal fistulas, or intra-abdominal abscesses 6 months prior to screening.
27. Currently pregnant, lactating or breastfeeding.
28. Required concomitant use of brivudine, sorivudine and analogues.
29. Required concomitant use of St John's Wort.
30. Required concomitant use of drugs known to prolong QT/QTc interval.
31. Required concomitant use of strong CYP3A4 inducers or strong CYP3A4 inhibitors. The use of strong CYP3A4 inducers within 2 weeks of first receipt of study drug or the use of strong CYP3A4 inhibitors within 1 week of first receipt of study drug is also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Oelmann, MD, PhD, Study Director — NuCana plc
Locations (59):
- United States (16):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Florida Health Medical Oncology - Davis Cancer Pavilion, Gainesville, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Morristown Medical Center, Morristown, New Jersey
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - USOR - Texas Oncology Northeast Texas, Tyler, Texas
  - Fred Hutchinson Cancer Center at Evergreen Health, Kirkland, Washington
  - Northwest Cancer Specialists, P.C. dba Compass Oncology - Vancouver Cancer Center, Vancouver, Washington
- France (9):
  - Strasbourg Oncology Liberale - Clinique Sainte-Anne, Strasbourg, Alsace
  - Hôpital Européen Marseille, Marseille, Bouches-du-Rhône
  - Centre Georges-François Leclerc, Dijon, Bourgogne-Franche-Comté
  - Centre Hospitalier Régional et Universitaire de Besançon - Hôpital Jean-Minjoz, Besançon, Doubs
  - Institut Bergonié, Bordeaux, Gironde
  - Centre Hospitalier Universitaire de Poitiers, Poitiers, Vienne
  - Centre Hospitalier UniversitaireNantes - Hôtel Dieu, Nantes
  - Hôpital Européen Georges-Pompidou, Paris, Île-de-France Region
  - Hôpital Foch, Suresnes, Île-de-France Region
- Germany (4):
  - München Klinik Neuperlach, München, Bavaria
  - Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Universitätsklinik Ulm - Oberen Eselsberg, Ulm, Tübingen
  - Charité Campus Virchow-Klinikum, Berlin
- Italy (8):
  - Azienda Ospedaliera Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Ospedale Santa Maria delle Croci di Ravenna, Faenza, Ravenna
  - Azienda Ospedaliero Universitaria Careggi, Florence, Tuscany
  - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Regionale San Carlo, Potenza
- Spain (14):
  - Institut Català d'Oncologia - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, La Coruña
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital de León, León
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (8):
  - Queen's Hospital, Romford, Essex
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - Royal Free London NHS Foundation Trust, London, Greater London
  - Guy's and Saint Thomas' NHS Foundation Trust, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Lancashire
  - Mount Vernon Cancer Centre - East and North Hertfordshire NHS Trust, Northwood, Middlesex
  - Velindre University NHS Trust, Cardiff
  - NHS Greater Glasgow and Clyde, Glasgow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 180 patients were randomized between April 2023 and August 2024
Groups:
- NUFIRI-bev Q1W: Arm A: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1, 8, 15, and 22.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. NUC-3373 1500 mg/m2 over 120 minutes on Days 1, 8, 15, and 22.
- NUFIRI-bev Q2W: Arm B: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1 and 15.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. NUC-3373 1500 mg/m2 over 120 minutes on Days 1 and 15
- FOLFIRI-bev Q2W: Arm C: Study treatment will be administered in 28-day cycles as follows:
  1. Bevacizumab 5 mg/kg on Days 1 and 15:
  2. LV 400 mg/m2 (or equivalent levo-LV) over 120 minutes on Days 1 and 15.
  3. Irinotecan 180 mg/m2 over 90 minutes (concurrently with the LV infusion) on Days 1 and 15.
  4. 5-FU 400 mg/m2 bolus on Days 1 and 15.
  5. 5-FU 2400 mg/m2 infusion over 46 hours on Days 1 and 15.
Period: Overall Study
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W
Started | 57 | 65 | 58
Completed | 35 | 34 | 32
Not Completed | 22 | 31 | 26
Not completed — Withdrawal by Subject | 2 | 0 | 5
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Progressive disease | 11 | 18 | 7
Not completed — No longer clinically benefitting | 2 | 1 | 0
Not completed — Sponsor decision | 5 | 9 | 8
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Patient non-compliance | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W | Total
Number analyzed (Participants) | 57 | 65 | 58 | 180
Age, Continuous [Median (Full Range); unit: Years] | 64.0 [38 to 78] | 64.0 [37 to 79] | 65.0 [27 to 85] | 64.0 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 27 | 24 | 72
  Male | 36 | 38 | 34 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 4 | 11
  White | 42 | 44 | 42 | 128
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 16 | 12 | 37
ECOG performance status [Count of Participants; unit: Participants] — The ECOG score describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The score runs from 0 to 5, with 0 denoting perfect health and 5 death. Patients with scores of 0 or 1 were eligible for this study:
  0 - Asymptomatic. Fully active, able to carry on all predisease activities without restriction
  1 - Symptomatic but completely ambulatory. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Participants
    0 | 31 | 36 | 38 | 105
    1 | 25 | 28 | 18 | 71
    Not reported | 1 | 1 | 2 | 4
Stage at initial diagnosis [Count of Participants; unit: Participants] — CRC is staged using the TNM system and grouped into Stages 0-4 (0-IV), with lower numbers indicating less advanced cancer.
  In Stages 1 and 2 (I and II), the cancer is confined to the bowel and has not spread to the lymph nodes or other organs.
  In Stage 3 (III), the cancer has spread to the lymph nodes but not to other organs.
  In Stage 4 (IV), the cancer has spread to distant parts of the body (e.g., the liver or lungs).
  Within each stage, subcategories show the extent of disease:
  A: Least advanced within that stage. B: More advanced than A. C: Most advanced within that stage.
  Participants
    Stage I (A-C) | 0 | 0 | 2 | 2
    Stage II (A-C) | 3 | 1 | 3 | 7
    Stage IIIA | 2 | 3 | 1 | 6
    Stage IIIB | 4 | 13 | 9 | 26
    Stage IIIC | 2 | 2 | 6 | 10
    Stage IV | 30 | 28 | 24 | 82
    Stage IVA | 11 | 8 | 9 | 28
    Stage IVB | 3 | 4 | 4 | 11
    Stage IVC | 1 | 3 | 0 | 4
    Not reported | 1 | 3 | 0 | 4
Primary tumor location [Count of Participants; unit: Participants]
  Colon - right side | 15 | 26 | 15 | 56
  Colon - left side | 20 | 23 | 21 | 64
  Colon - unknown | 6 | 5 | 8 | 19
  Rectum | 16 | 11 | 14 | 41
Liver metastases [Count of Participants; unit: Participants]
  Yes | 46 | 45 | 35 | 126
  No | 11 | 20 | 23 | 54
Number of metastatic sites [Count of Participants; unit: Participants]
  1 | 1 | 2 | 3 | 6
  2 | 9 | 10 | 7 | 26
  3 | 19 | 16 | 20 | 55
  4 or more | 28 | 36 | 28 | 92
  Not reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Progress-free Survival (PFS)
Description: PFS assessed according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1, defined as the time from randomisation to the first observation of objective tumour progression or death from any cause. Progression was defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in non-target lesions, or the appearance of new lesions.
Time Frame: Assessed from baseline to 30 days after last dose of study drug, up to 16 months
Measure: Median (Full Range); unit: Months
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W
Number analyzed (Participants) | 57 | 65 | 58
Months | 5.68 [0.03 to 11.17] | 5.52 [0.03 to 10.84] | 9.03 [0.03 to 15.01]

2. Secondary Outcome: Number of Patients Achieving a Reduction in Tumour Volume
Description: Objective response rate, defined as the percentage of patients achieving a complete (CR) or partial response (PR) to treatment. Response was measured by MRI scan and assessed per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria:
  CR= disappearance of all target lesions PR= at least a 30% decrease in the sum of the longest diameter of target lesions
Time Frame: Assessed from baseline to 30 days after last dose of study drug, up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W
Number analyzed (Participants) | 57 | 65 | 58
Participants | 4 | 12 | 12

3. Secondary Outcome: Number of Patients Achieving Disease Control
Description: Disease control rate, defined as the number of patients achieving a response (CR or PR) or stable disease (SD) as their best overall response. Disease control was measured by MRI scan and assessed using Response Evaluation Criteria in Solid Tumors (RECIST v1.1) criteria:
  CR= disappearance of all target lesions PR= at least a 30% decrease in the sum of the longest diameter of target lesions SD= neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease
Time Frame: Assessed from baseline to 30 days after last dose of study drug, up to 16 months
Measure: Count of Participants; unit: Participants
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W
Number analyzed (Participants) | 57 | 65 | 58
Participants | 35 | 42 | 46

ADVERSE EVENTS:
Time Frame: Each patient was assessed for adverse events from the date of informed consent until 30 days after the last dose of study treatment, up to 16 months.
Description: Adverse events and all-cause mortality were assessed in the safety population of patients who received at least one dose of study treatment. Compared to the participant flow numbers, there is one less patient per arm in the safety population as one patient per arm did not receive any study treatment.
Arm/Group | NUFIRI-bev Q1W | NUFIRI-bev Q2W | FOLFIRI-bev Q2W
All-Cause Mortality (participants affected / at risk) | 18/56 | 14/64 | 6/57
Serious Adverse Events (participants affected / at risk) | 11/56 | 13/64 | 17/57
Other Adverse Events (participants affected / at risk) | 55/56 | 62/64 | 57/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NUFIRI-bev Q1W (N=56) | NUFIRI-bev Q2W (N=64) | FOLFIRI-bev Q2W (N=57)
Hepatobiliary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1)
Inadequate analgesia (General disorders) | 1 (2) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion-related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Abdominal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Perihepatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NUFIRI-bev Q1W (N=56) | NUFIRI-bev Q2W (N=64) | FOLFIRI-bev Q2W (N=57)
Hypertension (Vascular disorders) | 5 (12) | 11 (13) | 8 (12)
Asthenia (General disorders) | 25 (45) | 23 (56) | 26 (60)
Fatigue (General disorders) | 10 (14) | 14 (23) | 11 (18)
Pyrexia (General disorders) | 9 (12) | 9 (10) | 5 (5)
Mucosal inflammation (General disorders) | 5 (8) | 3 (3) | 9 (13)
Influenza-like illness (General disorders) | 1 (2) | 1 (1) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 7 (8) | 7 (7)
Cough (General disorders) | 7 (7) | 6 (6) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3) | 4 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (6) | 5 (5) | 7 (8)
Alanine aminotransferase increased (Investigations) | 14 (46) | 4 (4) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 10 (32) | 4 (5) | 5 (5)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 7 (7) | 5 (6)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 11 (18)
Weight decreased (Investigations) | 4 (6) | 1 (1) | 5 (6)
Blood bilirubin increased (Investigations) | 4 (4) | 2 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 2 (5) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 1 (1) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 3 (5)
Infusion-related reaction (Injury, poisoning and procedural complications) | 4 (4) | 3 (4) | 0 (0)
Headache (Nervous system disorders) | 13 (25) | 6 (6) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (3) | 2 (3) | 6 (6)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 4 (5) | 2 (3)
Dizziness (Nervous system disorders) | 2 (5) | 4 (8) | 2 (2)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 4 (6) | 16 (28)
Anemia (Blood and lymphatic system disorders) | 7 (8) | 9 (16) | 5 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (7) | 3 (7) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 35 (113) | 33 (79) | 28 (76)
Nausea (Gastrointestinal disorders) | 29 (81) | 37 (80) | 22 (51)
Vomiting (Gastrointestinal disorders) | 22 (40) | 18 (41) | 9 (30)
Abdominal pain (Gastrointestinal disorders) | 18 (30) | 13 (22) | 8 (8)
Constipation (Gastrointestinal disorders) | 13 (21) | 7 (14) | 13 (19)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 6 (10) | 12 (23)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 5 (7) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 4 (11) | 5 (5) | 4 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 2 (2) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 4 (4) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 3 (4) | 2 (3) | 1 (1)
Salivary hypersecretion (Gastrointestinal disorders) | 3 (5) | 3 (3) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 3 (6) | 2 (2) | 0 (0)
Hypertransaminasemia (Hepatobiliary disorders) | 4 (11) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 14 (16)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12) | 4 (5) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (9) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 4 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (5) | 1 (1) | 3 (3)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 13 (18) | 11 (20) | 16 (22)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 4 (5) | 3 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5) | 1 (2) | 1 (3)

LIMITATIONS AND CAVEATS:
Due to the early closure of the study, many patients were censored for the efficacy endpoints and the data should therefore be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT05678257/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT05678257/SAP_001.pdf